CLINICAL TRIAL: NCT07208240
Title: Tb-PSMA-I&T Radionuclide Neo-Adjuvant Treatment in Patients With Locally Advanced Prostate Cancer Before Radical Prostatectomy: TbeforePROST Trial.
Brief Title: Tb-PSMA-I&T Radionuclide Before Radical Prostatectomy in Patients With Locally Advanced Prostate Cancer - TbeforePROST Trial.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, golan shay, Pro Shay Golan , Chair of Urology at Rabin Medical Cener, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC 833-23
Record Dates: First submitted 2025-08-12; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: High Risk Prostate Cancer
Keywords: High risk Prostate cancer; Radical Prostatectomy; PSMA; Theranostics; radionuclide therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving Tb-PSMA before RAdical prostatectomy (Experimental): Patients with high-risk locally advanced prostate cancer will receive 3 Tb-161-PSMA treatments followed by radical prostatectomy.
  Interventions: Drug: Tb-PSMA-I&T (Tb-PSMA)

INTERVENTIONS:
Drug: Tb-PSMA-I&T (Tb-PSMA) — Terbium-161 produce beta emission with the addition of Auger electrons which have higher linear energy transfer and a very short range. By that it has the potential to improve local and distal (micro-metastatic disease) efficacy with a similar safety profile. It will be given to patients with high risk locally advanced prostate cancer prior to Radical prostatectomy
  Other Names: radical prostatectomy

SUMMARY:
This is a multi-disciplinary collaboration between urologists, oncologists and nuclear medicine physicians from Beilinson hospital at Rabin Medical Center to address the major therapeutic challenge of locally advanced prostate cancer. Our aim is to evaluate the use of a novel treatment (Tb-PSMA) prior to the surgical removal of the prostate. This treatment has already shown initial promising results in patients with metastatic prostate cancer but has never been tested for locally advanced disease before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 years and older.
* Patients with high-risk localized prostate cancer (cT3/4 and/or Gleason score ≥ eight and/or prostate biopsy or PSA ≥ 20 ng/dl)
* High PSMA expression was confirmed according to PROMISE V2 8
* Patients should have an Eastern Cooperative Oncology Group (ECOG) performance status score of 1 or lower and a life expectancy of > 10 years.

Exclusion Criteria:

* Platelet count lower than 150×103/µl
* white blood cell count lower than 4×103/µl,
* haemoglobin concentration lower than 12mg/dl.
* albumin concentration lower than 3.5 g/dl.
* glomerular filtration rate (GFR) lower than 40 mL/min.
* usage of nephrotoxic drugs
* distant metastatic disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2028-08-12 (Estimated); Study Completion 2028-08-12 (Estimated)

PRIMARY OUTCOMES:
Number of Tb-PSMA adverse effects measured by CTCAE v4.0 and number of surgical complications - measured by the Clavien-Dindo Classification (2009) | 1 year
Surgical and clinical safety | 1 year
  The primary outcome is the safety of administering Tb-PSMA before radical prostatectomy, its impact on intra- and post-operative clinical course according to the Clavien-Dindo Classification.

SECONDARY OUTCOMES:
Immediate oncological outcomes as measured by number of patients with positive surgical margins and number of patients who achieved biochemical complete response | 3 months
  Secondary outcomes include the immediate response to treatment in terms of biochemical response. A post-surgical prostate specific antigen above 0.1 ng/ml is considered biochemical failure.

CONTACTS AND LOCATIONS:
Overall Officials: Shay Golan, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Beilinson Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided